CLINICAL TRIAL: NCT04879459
Title: Impact on Diagnostic Accuracy of Clinical Ultrasound Practical Teaching Exclusively Using Normal Gallbladder Patterns, a Pilot Double Blind Randomized Control Trial
Brief Title: Impact on Diagnostic Accuracy of a Specific Clinical Ultrasound Practical Teaching
Acronym: RCTpCUS
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: CUS gallbladder
Record Dates: First submitted 2021-04-26; First posted 2021-05-10 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Gallstone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group IG: The IG is constituted of participants, naïve to ultrasound use. Participants undergo a web-based video learning about gallbladder evaluation using CUS on day 0 (same video as in CG). Participants undertake 3 times a one-day CUS course consisting in 2 practical sessions of 10 times 10 minutes on 10 healthy volunteers on day 0, day 7 and day 10. One practical session takes place before lunchtime, the second one after lunchtime.
  Participants of IG don't have any contact with CG during study days. An evaluation is organized on day 60 to evaluate primary and secondary endpoints.
  Interventions: Other: Practical sessions to learn CUS exclusively on volunteers presenting a healthy gallbladder
- Control Group CG: The CG is constituted of participants, naïve to ultrasound use. Participants undergo a web-based video learning about gallbladder evaluation using CUS on day 0. Participants of CG undertake 2 practical CUS sessions of 10 times 10 minutes on 10 volunteers, at least 50% of them suffering from gallstones on day 0, day 7 and day 10. One session takes place before lunchtime, the second one after lunchtime.
  Participants of CG don't have any contact with IG during study days. An evaluation is organized on day 60 to evaluate primary and secondary endpoints.

INTERVENTIONS:
Other: Practical sessions to learn CUS exclusively on volunteers presenting a healthy gallbladder — The study days are 1 day apart for CG and IG but follow the exact same organization. Studytake place on day 0-10-30 (+/-2days). Practical sessions to learn CUS are organized either on volunteers presenting a healthy gallbladder or a pathological gallbladder (sludge, gallstones) (CG), either exclusively on volunteers presenting a healthy gallbladder (IG).
  Groups: Intervention Group IG

SUMMARY:
This research proposal is a pilot double-blind randomized control trial evaluating the impact on diagnostic accuracy of a Clinical UltraSound (CUS) teaching for gallbladder assessment using exclusively healthy volunteers for practical sessions. Classically, a number of 25 to 50 CUS of the gallbladder is reported to achieve competency. Many CUS curricula or guidelines recommend reporting pathological cases, either a certain amount, either generically, in their core-ultrasound competency requirements. Using healthy volunteers is rarely meant to verify the hypothesis that practical sessions based on exclusively normal patterns combined with presentation of pathological ultrasound loops or images during theoretical sessions, could further allow reaching diagnostic accuracy requirements in clinical practice. In the present study, participants will be medical students in their 5th year, naïve to CUS use. Participants will be randomly be distributed between a control group undergoing a standard practical teaching on models presenting uncomplicated gallstones or normal gallbladder (no gallstones), and an intervention group undergoing a practical teaching exclusively on models presenting a normal gallbladder. Participants will be "blinded" to study endpoints as well as to group allocation. After three days of practical teaching on day 0-10-30, students will be evaluated on day 60 by 2 external investigators blinded to students group allocation. Diagnostic accuracy for gallstones will be measured using sensitivity and specificity. Statistical analysis will be performed blinded to students' name using IBM SPSS statistics 26.0 (SPSS Inc., Chicago, IL, USA). As is classical, the statistical tests will be rejected whenever the observed p-value is smaller than 0.05. Corrections for multiple testing will be used. A comparable diagnostic accuracy between groups could further support the use of healthy volunteers during practical teaching and ease clinical ultrasound curricula. Such a finding wouldn't however carry away the need for enhancing competencies during clinical practice or the need for continuing medical education, as for any medical procedure.

DETAILED DESCRIPTION:
Background Critical care and emergency medicine are both specialties covering all types of pathologies concerning multiple etiologies and systems. Clinical UltraSound (CUS) curricula concerning those specialties are accordingly covering a wide range of ultrasound improved clinical examination. Recently, a questionnaire sent to American medical schools, reporting 84% response rate, enlightened that 55% of the clinical ultrasound course directors are emergency physicians. This supports the great implication of emergency medicine in CUS development.

In 2015, the International Federation for Emergency Medicine (IFEM) Point of Care UltraSound (PoCUS) published an evidence-based consensus document for CUS curriculum based on national and international guidelines. Previously, the Council of Emergency Medicine Residency Director-Academy of Emergency Ultrasound (CORD-AEUS) consensus established guidelines to organize CUS training and assess resident competencies. To actual knowledge, although CUS training programs around the globe support the use of specific training to achieve CUS introduction in the emergency departments endorsing its use, there are still significant variations among proposed curricula. The training requirements are mostly described for core-ultrasound. Generally, core-ultrasound curricula encompass the skill acquisition of extended-Focused Assessment Sonography for Trauma (e-FAST), Aortic Aneurysm Assessment (AAA), basic cardiac and lung ultrasound and basic procedural ultrasound. Some include biliary and urinary tract assessment whereas others consider biliary and urinary tract assessment part of advanced CUS teaching. Most other specialties however focus their ultrasound teaching on the field of interest. For instance, urologists learn how to perform an ultrasound assessment of the urinary tract or the prostate whereas gastroenterologists focus their ultrasound ability on bowel and biliary.

Currently, based on emergency medicine requirements, the CUS training consist of an initial introduction followed by gaining experience throughout image acquisition, image interpretation and clinical integration and finally achieving competency. Different approaches and methods of teaching are available and often a combination of those is recommended in available curricula description. Many recommend reporting pathological CUS cases among ultrasound images compeeled in a logbook, either a certain amount (20% to 50%), either generically, in their core-ultrasound competency requirements. Although its benefit for emergency medicine clinical practice is substantial and evidence based, the introduction of CUS in emergency physicians' practice is evidently time consuming possibly due to theoretical and practical sessions requirements and assessments as well as bedside supervision. Several curricula recently included CUS to emergency medicine requirements program and more broadly to medical students' courses. This brings to a large number the need for CUS bedside teaching combined with other sources of competence achievement.

In an emergency clinical setting, the use of CUS for hepatobiliary assessment is mostly centered on inflammation and obstruction. Cholecystitis is known to be, from 95% to 99% of cases secondary to gallstones. Gallstones are accessible to CUS and, included in the clinical context, can strengthen the suspicion of cholecystitis. In a systematic review performed in 2011, the pooled estimates for sensitivity and specificity were 89.8% (95% confidence interval (CI) 86.4% to 92.5%) and 88.0% (95% CI 83.7% to 91.4%), respectively for gallstones detection using EUS. This is consistent with this finding being valuable for clinical practice. Although some studies supported the number to achieve agreement with expert for gallbladder assessment to be 25 to 50, a prospective study including 1837 patients from 1999 to 2006, reported the learning curve of emergency physicians for the evaluation of gallbladder is poorly influenced by the number of bedside examinations. Those considerations suggest other sources of competency achievement should be evaluated rather than the number of examinations itself.

Classically, initial CUS introduction uses short lectures combined with demonstration, "hands-on" skill teaching, simulation sessions, discussions, web-based learning and practical scanning on volunteers, models and patients. Occasionally, pathological models are difficult to find and bedside teaching, apart from clinical shift, is exclusively possible on volunteers presenting a normal pattern. This enlightens the need for studies evaluating the CUS training pathway using exclusively healthy volunteers compared to the use of pathological findings during practical sessions. This is strengthen by the introduction of CUS courses among medical schools. Indeed, unlike residents or physicians, medical students don't have as much possibility to access practical CUS training on patients presenting pathological patterns.

The following study is meant to give insights about the CUS skills acquisition to accurately diagnose gallstones using exclusively training on healthy volunteers after a standardized web based theoretical teaching about pathological and non-pathological gallbladder CUS. This could support the use of only healthy volunteers during practical sessions. The teaching of pathological images recognition could exclusively be done throughout theoretical sessions. Although this would neither avoid the need for enhancing competencies bedside, neither avoid continuous logging activity and regular CUS continuing medical education, this could secondary help CUS teaching by reducing the need for bedside supervision during clinical shifts. Indeed, to knowledge, bedside supervision is difficult to achieve in some emergency departments and CUS fellows have trouble to properly fill out a " logbook ". Organizing CUS teaching around normal pattern recognition associated to a theoretical course presenting pathological findings could lead to change CUS fellows' assessment. Those could be evaluated theoretically using pathological ultrasound images or loops and could be evaluated practically on healthy volunteers. This would avoid compelling a " logbook " which can arise some ethical discussion about patient consent and use of images even if the latter are classically anonymized.

According to scope literature review, no randomized control study has been published establishing the skills acquisition for gallstones findings. This study being a pilot one, it will allow to precise the feasibility of a proper randomized control trial and to evaluate sample size. This study could also be the starting point of randomized control trials concerning the teaching of other pathological findings such as free fluid, aortic aneurism, cardiac assessment, hydronephrosis.

The Main objectives to evaluate if CUS skills to diagnose gallstones can be acquired by 5th year medical students naïve to CUS use exclusively throughout practical sessions on healthy volunteers after a standardized theoretical teaching using a web-based passive video learning.

The Trial design is a pilot double-blind randomized control trial. 20 participants are randomly assigned to CG or IG using pre-defined blocks of 10 participants per group. Consolidation of knowledge and skills' acquisition for gallbladder evaluation using CUS take place during 3 teaching sessions (day 0-10-30) given by CUS instructors on volunteers. Evaluation of diagnostic accuracy (day 60) is performed at the end of the 2 months teaching period by two blinded examiners. The teaching is performed according to an expanding time interval as supported by a recent review.

Study members

--> Instructors Instructors are selected from the population of experts in CUS of the gallbladder in Belgium ; they are invited to participate via e-mail.

Each instructor receives a financial compensation for participating to the study.

Instructors are not blinded to participants' allocation. Instructors sign a "non-disclosure agreement" meaning they cannot give information to a third party during the entire duration of the study.

--> Volunteers Healthy volunteers are invited to participate by e-mail. Volunteers are selected using a web-based questionnaire asking for characteristics (age, sex, BMI).

Volunteers presenting a pathological gallbladder status (gallstones, sludge), are invited to participate throughout the consultation of surgery of the "Cliniques Universitaires Saint-Luc", before an elective surgery is planned.

Volunteers are paired for age (+/- 5 years) and BMI (+/- 1) between groups to avoid selection bias.

Volunteers are eligible if:

* Between 18 and 70 years old
* Signed consent for participation and "non-disclosure agreement" 1 obtained
* Underwent a formal ultrasound previous to the study day in order to confirm gallbladder status (gallstones or sludge yes/no), performed by a CUS expert independent from the study
* Do not have persistent abdominal pain or cholecystitis symptoms Volunteers are committed to "non-disclosure agreement" about their gallbladder status during their participation to the study, except in case of medical consultation for personal matter.

  * Examiners Two examiners, blinded to participant allocation, evaluate practical skills of participants for gallbladder assessment using CUS on day 60.

Examiners are international experts in CUS coming from United Kingdom.

ELIGIBILITY:
Participants are eligible if:

* They are in 5th year of medical school
* They are naïve to CUS use
* They are available to participate to the 4 given dates of the study (day 0-10-30-60)

Inclusion Criteria:

* ≥ 18 years of age
* 5th year medical students
* Considered naïve to CUS
* Signed consent and signed non-disclosure agreement obtained

Exclusion Criteria:

* Unable to use CUS due to a disability
* Prior CUS skills

  ∗ Secondary exclusion criteria
* Unable to use CUS due to a new disability
* Unable to complete the four study days
* Breach of "non disclosure agreement"

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students →Participants An e-mail invitation is send three times over a two weeks period for participants enrollment. Participants are selected among medical students in their 5th year (Master 2). If e-mail is not sufficient, participants are invited during a medical course given in Université Catholique de Louvain. Medical students are invited to answer to a questionnaire defining their CUS use status (naïve or not) to assess for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for gallstones according to practical teaching (IG or CG) | Each participants will be evaluated at day 60 during a session of 20 minutes using volunteers for clinical ultrasound of the gallbladder
  sensitivity and specificity for gallstones diagnosis

SECONDARY OUTCOMES:
Difference betweeen pre-test and post-test results | Each participants will be evaluated at day 60 during a session of 20 minutes using volunteers for clinical ultrasound of the gallbladder
  after watching a web based video teaching about clinical ultrasound of the gallbladder
Confidence index for gallstones' diagnosis between Control Group (CG) and Intervention Group (IG). | Each participants will be evaluated at day 60 during a session of 20 minutes using volunteers for clinical ultrasound of the gallbladder
  Likert scale (0 = not confident --> 5 = perfectly confident)
Time to get CUS image between CG and IG | Each participants will be evaluated at day 60 during a session of 20 minutes using volunteers for clinical ultrasound of the gallbladder
  Time to get the image
Quality of the image between CG and IG | Each participants will be evaluated at day 60 during a session of 20 minutes using volunteers for clinical ultrasound of the gallbladder
  Image considered as interpretable or not by examiner

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Vanpee, PhD, Study Chair — Institut de recherche santé et société
Locations (1):
- Cliniques universitaires saint luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Corresponding groups and names will be kept in a secured database of the trial centre. Except for study coordinator, no access to data will be possible for any other member of the study. A list of correspondence between study identification number and the other identifying data initially collected will be kept under the responsibility of the promoter. This list is kept for the statutory period of time provided for this type of research. The protection of the patient's personal data will be guaranteed according to the European General Data Protection Regulation of 27 April 2016 (in application since 25 May 2018), to the Belgian Law of 30 July 2018 on the protection of privacy with regard to the processing of personal data and to the Belgian Law of 22 August 2002 on the rights of the patient.

REFERENCES:
- [Background] American College of Emergency Physicians. American College of Emergency Physicians. ACEP emergency ultrasound guidelines-2001. Ann Emerg Med. 2001 Oct;38(4):470-81. No abstract available. PMID 11574810
- [Background] Ultrasound Guidelines: Emergency, Point-of-Care and Clinical Ultrasound Guidelines in Medicine. Ann Emerg Med. 2017 May;69(5):e27-e54. doi: 10.1016/j.annemergmed.2016.08.457. No abstract available. PMID 28442101
- [Background] Atkinson P, Bowra J, Lambert M, Lamprecht H, Noble V, Jarman B. International Federation for Emergency Medicine point of care ultrasound curriculum. CJEM. 2015 Mar;17(2):161-70. doi: 10.1017/cem.2015.8. PMID 26052968
- [Background] Back SJ, Darge K, Bedoya MA, Delgado J, Gorfu Y, Zewdneh D, Reid JR. Ultrasound Tutorials in Under 10 Minutes: Experience and Results. AJR Am J Roentgenol. 2016 Sep;207(3):653-60. doi: 10.2214/AJR.16.16402. Epub 2016 Jun 8. PMID 27276225
- [Background] Dinh VA, Lakoff D, Hess J, Bahner DP, Hoppmann R, Blaivas M, Pellerito JS, Abuhamad A, Khandelwal S. Medical Student Core Clinical Ultrasound Milestones: A Consensus Among Directors in the United States. J Ultrasound Med. 2016 Feb;35(2):421-34. doi: 10.7863/ultra.15.07080. Epub 2016 Jan 18. PMID 26782162
- [Background] Gaspari RJ, Dickman E, Blehar D. Learning curve of bedside ultrasound of the gallbladder. J Emerg Med. 2009 Jul;37(1):51-6. doi: 10.1016/j.jemermed.2007.10.070. Epub 2008 Apr 25. PMID 18439787
- [Background] Jain A, Mehta N, Secko M, Schechter J, Papanagnou D, Pandya S, Sinert R. History, Physical Examination, Laboratory Testing, and Emergency Department Ultrasonography for the Diagnosis of Acute Cholecystitis. Acad Emerg Med. 2017 Mar;24(3):281-297. doi: 10.1111/acem.13132. PMID 27862628
- [Background] Jang TB, Ruggeri W, Dyne P, Kaji AH. The learning curve of resident physicians using emergency ultrasonography for cholelithiasis and cholecystitis. Acad Emerg Med. 2010 Nov;17(11):1247-52. doi: 10.1111/j.1553-2712.2010.00909.x. PMID 21175524
- [Background] Lewis D, Rang L, Kim D, Robichaud L, Kwan C, Pham C, Shefrin A, Ritcey B, Atkinson P, Woo M, Jelic T, Dallaire G, Henneberry R, Turner J, Andani R, Demsey R, Olszynski P. Recommendations for the use of point-of-care ultrasound (POCUS) by emergency physicians in Canada. CJEM. 2019 Nov;21(6):721-726. doi: 10.1017/cem.2019.392. No abstract available. PMID 31771691
- [Background] Lewiss RE, Pearl M, Nomura JT, Baty G, Bengiamin R, Duprey K, Stone M, Theodoro D, Akhtar S. CORD-AEUS: consensus document for the emergency ultrasound milestone project. Acad Emerg Med. 2013 Jul;20(7):740-5. doi: 10.1111/acem.12164. PMID 23859589
- [Background] Mengel-Jorgensen T, Jensen MB. Variation in the use of point-of-care ultrasound in general practice in various European countries. Results of a survey among experts. Eur J Gen Pract. 2016 Dec;22(4):274-277. doi: 10.1080/13814788.2016.1211105. Epub 2016 Aug 3. PMID 27487159
- [Background] Olszynski P, Kim D, Chenkin J, Rang L. The core emergency ultrasound curriculum project: A report from the Curriculum Working Group of the CAEP Emergency Ultrasound Committee. CJEM. 2018 Mar;20(2):176-182. doi: 10.1017/cem.2017.44. Epub 2017 Jun 19. PMID 28625217
- [Background] Rempell JS, Saldana F, DiSalvo D, Kumar N, Stone MB, Chan W, Luz J, Noble VE, Liteplo A, Kimberly H, Kohler MJ. Pilot Point-of-Care Ultrasound Curriculum at Harvard Medical School: Early Experience. West J Emerg Med. 2016 Nov;17(6):734-740. doi: 10.5811/westjem.2016.8.31387. Epub 2016 Sep 12. PMID 27833681
- [Background] Ross M, Brown M, McLaughlin K, Atkinson P, Thompson J, Powelson S, Clark S, Lang E. Emergency physician-performed ultrasound to diagnose cholelithiasis: a systematic review. Acad Emerg Med. 2011 Mar;18(3):227-35. doi: 10.1111/j.1553-2712.2011.01012.x. PMID 21401784
- [Background] Salmon M, Landes M, Hunchak C, Paluku J, Malemo Kalisya L, Salmon C, Muller MM, Wachira B, Mangan J, Chhaganlal K, Kalanzi J, Azazh A, Berman S, Zied ES, Lamprecht H. Getting It Right the First Time: Defining Regionally Relevant Training Curricula and Provider Core Competencies for Point-of-Care Ultrasound Education on the African Continent. Ann Emerg Med. 2017 Feb;69(2):218-226. doi: 10.1016/j.annemergmed.2016.07.030. Epub 2016 Dec 11. PMID 27974170
- [Background] Villar J, Summers SM, Menchine MD, Fox JC, Wang R. The Absence of Gallstones on Point-of-Care Ultrasound Rules Out Acute Cholecystitis. J Emerg Med. 2015 Oct;49(4):475-80. doi: 10.1016/j.jemermed.2015.04.037. Epub 2015 Jul 7. PMID 26162764
- See also: Credentialing For Emergency Medicine Ultrasonography — https://acem.org.au/getmedia/ee68a734-7634-425d-865a-f5e17dc8b4e4/P733_Policy-on-Credentialing-for-Emergency-Medicine-Ultrasonography_v1_Aug-2019